CLINICAL TRIAL: NCT03951298
Title: International Tracking Neurodegeneration in Early Wolfram Syndrome
Brief Title: I-Tracking Neurodegeneration in Early Wolfram Syndrome
Acronym: I-TRACK
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201808060
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Wolfram Syndrome
Keywords: Diabetes Mellitus; Diabetes Insipidus; Optic Atrophy; Deafness
MeSH Terms: conditions — Wolfram Syndrome; Diabetes Mellitus; Diabetes Insipidus; Optic Atrophy; Deafness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Wolfram Syndrome Patients: Participant has confirmation of a WFS1 mutation OR Both of the following conditions: diabetes mellitus requiring insulin and optic nerve atrophy diagnosed by a physician. Both conditions diabetes mellitus and optic nerve atrophy had to be diagnosed at age younger than 18 years old
- Proxy Group: Adult Biological parent(s), biological caregiver or non-biological caregiver of adult and minor participants in the any of the groups.

SUMMARY:
Wolfram syndrome (WFS; OMIM #222300) is a rare autosomal recessive disease clinically defined in 1938 as the combination of childhood-onset insulin dependent diabetes, optic nerve atrophy, diabetes insipidus and deafness. Based on early descriptions, neurological features were thought to appear later in the disease with death occurring in middle adulthood. Importantly, the major causative gene (WFS1) was identified in 1998. This discovery allowed researchers to determine that the WFS1 gene encodes the protein wolframin, which helps protect cells from endoplasmic reticulum (ER) stress-mediated apoptosis, potentially via intracellular calcium homeostasis. Pathogenic mutations in WFS1 can result in death or dysfunction of cells that are under high ER stress, such as insulin-producing pancreatic β cells, causing insulin dependent diabetes. In addition, knowing the causative gene has allowed researchers to identify patients by their WFS1 mutation rather than the classic set of symptoms, leading to the increasing realization that the WFS1-related phenotype (including neurologic symptoms) is much more variable than previously understood. The first iteration of this grant (HD070855 "Tracking Neurodegeneration in Early Wolfram Syndrome") contributed to this shift in understanding. In this time, the research team has built a successful annual research clinic for WFS, that has met or exceeded recruitment goals for patients and controls, validated a clinical severity rating scale for WFS, described an unexpectedly early neurophenotype of reduced balance, smell identification and ventral pons volume, identified alterations in traditional diffusion tensor imaging (DTI) metrics that suggest hypomyelination as a pervasive neuropathological feature of WFS and provided justification for the selection of two primary outcomes (visual acuity and ventral pons volume) in a newly funded clinical efficacy study in WFS (Barrett, PI).

DETAILED DESCRIPTION:
In this new grant, researchers hypothesize that ER stress-related dysfunction could inhibit production of myelin during neurodevelopment in WFS, as active and developing oligodendrocytes (cells that produce myelin in the brain) are more vulnerable to ER stress than mature ones. However, standard DTI methods conflate inflammatory processes (which can also be associated with ER stress) in the extra-axonal space with metrics of axonal and myelin integrity, leading to potentially confounded measurements. The research team proposea to collect novel, validated diffusion sequences on a new state of the art MRI scanner (Siemens Prisma) and apply cutting-edge analysis approaches to measure white matter integrity throughout the brain and in the optic nerve, improving the ability to draw conclusions about axonal and myelin integrity over time. Researchers will assess WFS patients annually at our WU Wolfram Research Clinic using these methods.

Findings from this work may indicate future targets for brain-specific intervention, identify outcome measures or high-risk subgroups for clinical trials targeting neurological symptoms. These data will also greatly expand our understanding of the cross-sectional and longitudinal phenotype of WFS1-mutation related disorders, rather than classically defined Wolfram Syndrome. Such knowledge will have a significant impact on patients and families by allowing physicians to provide more accurate prognoses. Finally, forms of ER stress-mediated apoptosis have been implicated in more common neurodegenerative, endocrine and neurodevelopmental diseases, which may benefit from the insights gained here.

ELIGIBILITY:
Wolfram Syndrome Group (WFS):

Inclusion Criteria:

* Patient has confirmation of a WFS1 mutation OR
* Both of the following conditions:

  * diabetes mellitus requiring insulin and
  * optic nerve atrophy diagnosed by a physician.

Exclusion Criteria:

* Patient is unaware of their diagnosis.
* Inability of patient or guardian to understand informed consent.
* Advanced disease that makes traveling too problematic and/or uncomfortable for the patient and/or guardian, such as the use of a ventilator or inability to walk.

Sibling Group: Biological, half and step-siblings who do not have any symptoms of WFS and/or have had genetic testing to show that they do not have WFS may participate.

Exclusion Criteria:

• Inability of participant or guardian to understand informed consent.

Proxy Group: Adult Biological parent(s), biological caregiver, or non-biological caregiver of adult and minor participants in any of the four groups.

Inclusion criteria:

• Biological or non-biological parent/caregiver (proxy) of a participant.

Exclusion Criteria:

• Proxy is unaware of the participant's diagnosis (as it applies).

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Age, gender and handedness-matched participants between the age of 1 day to no upper limit.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in regional brain volumes over time | Annually for 5 years.
  MRI measures of regional brain volumes over time

SECONDARY OUTCOMES:
Change in disease severity score | Annually for 5 years.
  WURS physical severity score over time

CONTACTS AND LOCATIONS:
Overall Officials: Tamara G Hershey, PhD, Principal Investigator — Washington University Medical School
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States